CLINICAL TRIAL: NCT01903343
Title: Repeatability and Reproducibility of the Measurement of Young's Modulus Using Shear Wave Elastography in Volunteers
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: 2013AN01
Record Dates: First submitted 2013-07-11; First posted 2013-07-19 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Anesthesia
Keywords: Shear wave; Elastography; Repeatability and Reproducibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Single group of healthy male medical students at Ninewells Hospital & Medical School, Dundee.
  Interventions: Device: shear wave elastography

INTERVENTIONS:
Device: shear wave elastography — ultrasound

SUMMARY:
The aim of the study is to assess the accuracy of shear wave elastography in volunteers. Shear wave elastography is a non-invasive, non-painful measure of tissue stiffness obtained using an ultrasound machine. It may be easier to think of shear wave elastography as a special type of ultrasound imaging which gives doctors a colour picture of body structures based on their stiffness.

DETAILED DESCRIPTION:
Shear wave elastography is a quantitative ultrasound modality increasingly used to differentiate between "hard" breast cancer masses and "soft" normal tissue. Unlike strain elastography, shear wave elastography applies a non-compressive longitudinal acoustic radiation force to underlying tissues, inducing transverse shear waves. Studies in Thiel embalmed human cadavers have shown significant differences in Young's modulus between intraneural and extraneural tissue, and ready colour differentiation between tissues.

Therefore, before clinical application, we wish to measure the repeatability and reproducibility of Young's modulus of intraneural and extraneural tissue in volunteers. For measurement, a region of interest (ROI) will be selected over the appropriate nerve and adjacent tissue. The ROI results will be regarded as paired data. Paired data will be measured over and adjacent to the interscalene C5 nerve root, infraclavicular lateral cord, musculocutaneous, median, femoral, saphenous and sciatic nerves.

ELIGIBILITY:
Inclusion Criteria:

* Fit healthy male volunteers between 18 and 35 years of age.
* Participants with an ASA score of 1.
* Capacity to provide informed consent.

Exclusion Criteria:

* All females.
* Male participants aged <18 years and >35 years of age.
* ASA score 2 or above.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study of 8 subjects - volunteer medical students. Recruitment: Male medical students at Ninewells Hospital & Medical School, Dundee.
  Male medical students will be e-mailed by the chief investigator.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To determine the reproducibility of Young's modulus in volunteers using shear wave elastography | 4 hours
  To determine the reproducibility of Young's modulus in volunteers using shear wave elastography
To determine the repeatability Young's modulus in volunteers using shear wave elastography | 4 hours
  To determine the repeatability Young's modulus in volunteers using shear wave elastography

SECONDARY OUTCOMES:
Video Young's Modulus | max 2 minutes
  To video changes in tissue stiffness (using the elastography colour map) in concert with changes in the B-Mode image

CONTACTS AND LOCATIONS:
Overall Officials: Graeme A McLeod, MBChB FRCA, Principal Investigator — NHS Tayside
Locations (1):
- Department of Anaesthesia, Ninewells Hospital & Medical School, Dundee, United Kingdom

REFERENCES:
- [Background] Macfarlane AJ, Prasad GA, Chan VW, Brull R. Does regional anesthesia improve outcome after total knee arthroplasty? Clin Orthop Relat Res. 2009 Sep;467(9):2379-402. doi: 10.1007/s11999-008-0666-9. Epub 2009 Jan 7. PMID 19130163
- [Background] Evans A, Whelehan P, Thomson K, McLean D, Brauer K, Purdie C, Jordan L, Baker L, Thompson A. Quantitative shear wave ultrasound elastography: initial experience in solid breast masses. Breast Cancer Res. 2010;12(6):R104. doi: 10.1186/bcr2787. Epub 2010 Dec 1. PMID 21122101
- [Background] Liu SS, YaDeau JT, Shaw PM, Wilfred S, Shetty T, Gordon M. Incidence of unintentional intraneural injection and postoperative neurological complications with ultrasound-guided interscalene and supraclavicular nerve blocks. Anaesthesia. 2011 Mar;66(3):168-74. doi: 10.1111/j.1365-2044.2011.06619.x. PMID 21320084
- [Background] Neal JM. Ultrasound-guided regional anesthesia and patient safety: An evidence-based analysis. Reg Anesth Pain Med. 2010 Mar-Apr;35(2 Suppl):S59-67. doi: 10.1097/AAP.0b013e3181ccbc96. PMID 20216027
- [Background] Neal JM, Brull R, Chan VW, Grant SA, Horn JL, Liu SS, McCartney CJ, Narouze SN, Perlas A, Salinas FV, Sites BD, Tsui BC. The ASRA evidence-based medicine assessment of ultrasound-guided regional anesthesia and pain medicine: Executive summary. Reg Anesth Pain Med. 2010 Mar-Apr;35(2 Suppl):S1-9. doi: 10.1097/AAP.0b013e3181d22fe0. PMID 20216019